CLINICAL TRIAL: NCT06500949
Title: Effects of Vagus Nerve Pulmonary Branch Block on Postoperative Cough After Thoracoscopic Lung Resection
Brief Title: Effects of Vagus Nerve Pulmonary Branch Block on Postoperative Cough After VATS Lung Resection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024-0618
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-06

CONDITIONS: Postoperative Cough; Thoracoscopy; Pulmonary Resection; Vagus; Nerve Block
Keywords: Chronic cough; Postoperative cough; Thoracoscopy or Video-assisted thoracoscopic surgery; Pulmonary resection or Lung resection; Vagus
MeSH Terms: conditions — Chronic Cough

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vagus nerve pulmonary branch block group (V group) (Experimental): After thoracotomy, under direct thoracoscopic visualization, 2.5 ml of 0.375% ropivacaine was injected in proximity to the main trunk of the pulmonary branches of the vagus nerve.
  Interventions: Procedure: Vagus Nerve Pulmonary Branch Block
- Control group (C group) (Placebo Comparator): After thoracotomy, under direct thoracoscopic visualization, 2.5 ml of normal saline was administered in the vicinity of the principal trunk of the pulmonary branches of the vagus nerve.
  Interventions: Procedure: Vagus Nerve Pulmonary Branch Injection

INTERVENTIONS:
Procedure: Vagus Nerve Pulmonary Branch Block — Following thoracotomy, the thoracic surgeon, under direct thoracoscopic guidance, used forceps to elevate the apex of the lung, thus exposing the main trunk of the pulmonary branches of the vagus nerve. The injection needle was then advanced from a lateral-to-medial direction, and 2.5 ml of 0.375% ropivacaine was administered in close proximity to the targeted vagal branch.
  Arms: Vagus nerve pulmonary branch block group (V group)
Procedure: Vagus Nerve Pulmonary Branch Injection — Following thoracotomy, the thoracic surgeon, under direct thoracoscopic guidance, used forceps to elevate the apex of the lung, thus exposing the main trunk of the pulmonary branches of the vagus nerve. The injection needle was then advanced from a lateral-to-medial direction, and 2.5 ml of normal saline was administered in close proximity to the targeted vagal branch.
  Arms: Control group (C group)

SUMMARY:
Postoperative cough after pulmonary resection is a common issue seen after thoracic surgeries, hindering patients' recovery and affecting their postoperative quality of life. While vagus nerve pulmonary branch block has been known to reduce intraoperative coughing, its impact on postoperative cough post lung resection is uncertain. This study aims to assess the effects of vagus nerve pulmonary branch block on postoperative cough after VATS lung resection. A randomized controlled trial involving 104 thoracoscopic lung resection patients will assign them randomly to a vagus nerve pulmonary branch block group or a control group. The primary outcome measure is the postoperative cough incidence 3 weeks after lung resection. The secondary outcomes include assessing hoarseness in PACU, peak expiratory flow (PEF) on the first post-op day, NRS scores for cough, and LCQ-MC scores at 3 weeks post-surgery, as well as cough occurrence, NRS scores, and LCQ-MC scores at 8 weeks post-procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years old.
* BMI between 18 and 30 kilograms per square meter (kg/m²).
* ASA Physical Status Classification of I, II, or III.
* Preoperative pulmonary imaging demonstrating peripheral lesions, with clinical staging T≤2, N≤1, M0.
* Undergone thoracoscopic lung resection surgery.
* Patients managed by the same lead surgeon's team.
* Obtained informed consent, with patients agreeing and signing the informed consent document.

Exclusion Criteria:

* Patients with a history of chemotherapy or previous pulmonary surgery.
* Presence of chronic cough due to respiratory infectious diseases, pharyngitis, rhinitis, COPD, asthma, post-nasal drip syndrome, etc.
* Individuals exhibiting ECG abnormalities such as atrial fibrillation, bundle branch block, frequent ventricular premature beats, pre-excitation syndrome, etc.
* Currently using ACE inhibitor medications.
* Presence of preoperative hoarseness.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative cough following lung resection at 3 weeks post-operation | at 3 weeks post-operation
  The incidence of post-lung resection cough was assessed at 3 weeks postoperatively.

SECONDARY OUTCOMES:
Condition of hoarseness in PACU | during in PACU, an average of 1 hour
  Assessment of hoarseness in PACU following surgery
Peak expiratory flow rate on postoperative day 1 | on postoperative day 1
  Measurement of peak expiratory flow on postoperative day 1
Numerical Rating Scale for cough intensity at 3 weeks post-operation | at 3 weeks post-operation
  The scale ranges from 0 to 10, with 0 indicating no cough and 10 representing the worst imaginable cough.Higher scores on the Numerical Rating Scale for cough intensity indicate a more severe cough condition.
Leicester Cough Questionnaire for Measuring Chronic Cough at 3 weeks post-operation | at 3 weeks post-operation
  The LCQ-MC score ranges from a minimum of 0 to a maximum of 21, with three dimensions: physical, psychological, and social. Each dimension is scored from 1 to 7, and the total score is the sum of the three dimensions.Higher scores on the LCQ-MC indicate better health-related quality of life. A score of 0 represents the worst possible quality of life, while a score of 21 represents the best possible quality of life in relation to cough.
Incidence of postoperative cough following lung resection at 8 weeks post-operation | at 8 weeks post-operation
  The incidence of post-lung resection cough was assessed at 8 weeks postoperatively.
Numerical Rating Scale for cough intensity at 8 weeks post-operation | at 8 weeks post-operation
  The scale ranges from 0 to 10, with 0 indicating no cough and 10 representing the worst imaginable cough.Higher scores on the Numerical Rating Scale for cough intensity indicate a more severe cough condition.
Leicester Cough Questionnaire for Measuring Chronic Cough at 8 weeks post-operation | at 8 weeks post-operation
  The LCQ-MC score ranges from a minimum of 0 to a maximum of 21, with three dimensions: physical, psychological, and social. Each dimension is scored from 1 to 7, and the total score is the sum of the three dimensions.Higher scores on the LCQ-MC indicate better health-related quality of life. A score of 0 represents the worst possible quality of life, while a score of 21 represents the best possible quality of life in relation to cough.

CONTACTS AND LOCATIONS:
Locations (1):
- Second affiliated Hospital School of Medicine,Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No